CLINICAL TRIAL: NCT00537888
Title: Diagnosis of Pulmonary Candidiasis
Brief Title: Clinical Significance of Smear or Culture Positive for Candida Spp. From Sputum Three Times a Week
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Capital Medical University, Beijing Chaoyang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CYH-CMU
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2009-07

CONDITIONS: Pulmonary Candidiasis
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fluconazole — Intravenous or oral 400 md/d

SUMMARY:
The definition of pulmonary candidiasis is still unclear.In China, isolation of candida spp. form sputum twice or three times a week has been regarded as the microbiological evidence of pulmonary candidiasis. The investigators hypothesize that patients who present respiratory symptoms and lung infiltrates together with smear of culture positive for candida spp. from sputum three times a week can not be diagnosed as pulmonary candidiasis.

ELIGIBILITY:
Inclusion Criteria:

* 85ys>age>14ys
* APACHE II<25
* Lung infiltrates together with at least one of the following symptoms:cough, sputum, dyspnea with or without fever
* smear or culture positive for candida spp. from sputum

Exclusion Criteria:

* Pregnancy
* Hypersensitivity to fluconazole
* Isolated candida was non-sensitive to fluconazole
* Severe liver or renal diseases who can not tolerate fluconazole treatment
* With at least one of the following high risk factors:organ transplantation, neutropenia>10ds, long term glucocorticoids therapy(equal to prednisone 30mg/d longer than 2 weeks), immunosuppressive therapy within 30ds, AIDS
* With one of the microbiological evidence:isolation of candida spp. from blood or other kinds of sterile site(not including urine), filamentous fungi isolated from sputum or BALF, cryptococcus isolated from sputum or CSF, galactomannan antigen positive twice for blood
* Probable or possible pulmonary aspergillosis
* Definite oral or esophageal candidiasis

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
invasive candidiasis | in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cao, Doctor, Principal Investigator — Beijing Chaoyang Hospital, Affiliate of Capital Medical University
Locations (1):
- Beijing Chaoyang Hospital,Affiliate of Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Cao B, Cai BQ, Wang H, Zhou CY, Wang P, Liu HR, Zhang H, Xu L, Xu KF, Xu WB, Zhu YJ, Li XG. [A study of 152 cases of pulmonary fungal infection: reevaluation of the microbiological spectra]. Zhonghua Jie He He Hu Xi Za Zhi. 2007 Apr;30(4):279-83. Chinese. PMID 17651612